CLINICAL TRIAL: NCT05837546
Title: Neurodynamic of the Human Brain Underlying Animal-assisted Intervention in Healthy Adults
Acronym: NMAAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Karin Hediger (Other)
Responsible Party: Sponsor-Investigator, Dr. Karin Hediger, Professor, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-00206
Record Dates: First submitted 2023-03-21; First posted 2023-05-01 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Animal-assisted Intervention

STUDY DESIGN:
Intervention Model Description: within-subject randomized controlled trial with repeated measurement
Masking Description: Due to the nature of the conditions, the experimenters and the participants cannot be blinded as it is obvious if the animal is present or not. Nevertheless, participants will not be informed of the order of the conditions before the beginning of the measurement and to minimize bias they will not be informed about our hypotheses and that we are interested in the effects of the presence of a dog.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Real dog (Experimental): presence of a real dog, contact with participant for 5 minutes
  Interventions: Other: Animal-assisted intervention
- replica dog (Active Comparator): presence of a replica dog, contact with participant for 5 minutes
  Interventions: Other: Factice dog intervention
- plant (Active Comparator): presence of a plant, contact with participant for 5 minutes
  Interventions: Other: Plant intervention

INTERVENTIONS:
Other: Animal-assisted intervention — presence of a dog, contact between dog and participant
  Arms: Real dog
Other: Factice dog intervention — presence of a factice dog, contact between factice dog and participant
  Arms: replica dog
Other: Plant intervention — presence of a plant, contact between plant and participant
  Arms: plant

SUMMARY:
The electrical activity of the brain will be studied using EEG on healthy young adults. The frontal alpha asymmetry (FAA) of the participant will be measured during three conditions: presence of a dog, presence of a replica dog, presence of a plant. The researchers hypothesize that the activity in the left frontal hemisphere is greater than in the right during an animal-assisted intervention compared to the control conditions.

DETAILED DESCRIPTION:
The primary objective of this study is to measure the alpha power spectrum of an electroencephalogram measurements in the prefrontal cortex of healthy adults during an AAI. The investigators aim to measure established biomarkers of motivation and positive emotions in the EEG recordings and associate them with the AAI. The investigators will use three pair of electrodes to focus on the frontal and prefrontal cortex: F3-F4/F7-F8 and Fp1-Fp1 according to the international 10-20 system to calculate three FAAs. The study is a within-subject randomized controlled trial with repeated measurement. All participants are assigned to the same procedures: Each participant will have 3 measurements in 3 independent sessions. In each session the participants are exposed to 3 conditions (in total participant are exposed 3 times to each condition, once per session). The order of the exposition is randomized for every session. The intervention is an animal-assisted intervention. Usually, an animal is involved in a treatment with the aim of enhancing a therapeutic aim. In our study, there is no therapeutic setting but rather just the presence of a dog. The investigators describe "presence" by, whenever possible, a physical contact between the dog and the participant. This contact will be established by instructing the dog to lie down next to the participant and by instructing the participant to gently pet the dog. This contact cannot be guaranteed during the whole duration of the measurement because the dog is a living creature and will not be forced to do anything against its will.

As control conditions the investigators use a replica therapy dog (Joy for All) and a condition with no dog but the presence of a plant. The plant was chosen as to control for the mere presence and engagement with an object and because the impact of the presence of a plant in the frontal brain electrical activity has been studied before. In both control conditions, the intervention will be as similar as possible to the real dog condition with a physical contact between the object and the participants.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent as documented by signature
* Age ≥ 18 years

Exclusion Criteria:

* Fear of or allergies to dogs (self-reported)
* Any acute or chronic disease (e.g. chronic pain, hypertension, heart disease, renal disease, liver disease, diabetes)
* Current medications (e.g. psychoactive medication, narcotics, intake of analgesics) or being currently in psychological or psychiatric treatment
* Current or regular drug consumption (THC (24h before visit), cocaine, heroin, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
frontal alpha asymmetry (FAA) | 3 times + baseline per sessions, 1 hours per week, for 3 weeks
  difference between right and left hemispheres of the log transformed values of the averaged alpha power: (ln[right]-ln[left])

SECONDARY OUTCOMES:
Intrinsic Motivation Index (IMI) | 3 times per sessions, 1 hours per week, for 3 weeks
  questionnaire reporting motivation after a task
"Multidimensional well-being questionnaire" (MDWBQ) | 3 times + baseline per sessions, 1 hours per week, for 3 weeks
  questionnaire reporting general state of mind

CONTACTS AND LOCATIONS:
Locations (1):
- University of Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided